CLINICAL TRIAL: NCT01000740
Title: An International Expanded Access Clinical Programme With ZD1839 (IRESSATM) for Patients With Advanced Non-small Cell Lung Cancer (NSCLC) China Amendment 1: A Study on the Long Term Survivals in an Expand Access Program (EAP) of Iressa
Brief Title: A Study on the Long Term Survivals in an Expand Access Program (EAP) of Iressa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0052 SubStudy
Record Dates: First submitted 2009-09-07; First posted 2009-10-23 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EAP; Long term survival (3 years); Gefitinib; efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Long term survivors who has been used IRESSA for more than 3 years and are still on gefitinib treatment
  Interventions: Genetic: EGFR Mutation Test; Genetic: Ki-67 protein expression
- 2 (No Intervention): Long term survivors who has been used IRESSA for more than 3 years but have already terminated from EAP
- 3 (No Intervention): Fast-progressors who defined as no more than 1 follow-up visit after recruitment with the reason of discontinuation being

INTERVENTIONS:
Genetic: EGFR Mutation Test — Explore the EGFR mutation status from both tumour tissue sample and the free DNA in the peripheral blood using appropriate method(s) which may include ARMS assay, ME-PCR coupled sequencing and regular sequencing.
  Arms: 1
Genetic: Ki-67 protein expression — Ki-67 protein expression in tissue will be analysed by IHC method.
  Arms: 1

SUMMARY:
The primary objective is to describe the quality of life of long-term survivors who are not terminated from the EAP.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Participated in the Iressa EAP in China.
* Diagnosed as NSCLC.
* Patients who started EAP at least 3 years before this study initiated and have not yet terminated from the EAP (active long-term survivors).
* Patients who consent to provide blood sample and available archival tumour tissue sample for EGFR gene testing (provision of tumour tissue sample is optional).

Exclusion Criteria:

* Patients who disagree to participate this study.
* Patients in whose medical objection was recorded to use the existing data from medical practice for scientific research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Describe the quality of life of long-term survivors who are not terminated from the EAP

SECONDARY OUTCOMES:
To describe the current tumour control status via RECIST
To collect the risk factors related to prognosis in addition to the information already collected from EAP (age, gender, histology, smoking history, previous history of anti-cancer treatment, disease stage before starting gefitinib treatment, etc.)
To describe the treatment compliance of gefitinib in these patients
To describe the current clinical status of long-term survivors in the EAP program by clinical
To compare the key clinical features (age group, gender, histology, smoking history, disease stage, treatment-naive or pre-treated, response to prior chemotherapy,) in fast-progressors versus long-term survivals.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Atkin, Study Director — AstraZeneca; Louis Zhang, Study Chair — AstraZeneca; Longyun Li, Principal Investigator — Peking Union Medical College Hospital
Locations (9):
- China (9):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Li L, Zhong W, Liao M, Chen L, Han B, Guan Z, Yu S, Liu X, Wu Y, Jiang G, Xu J, Chen J, Tao M, Luo R, Li W, Xu N, Zhao X, Wang M. [A study on the long-term non-small cell lung cancer survivors in the Expand Access Program of gefitinib in China]. Zhongguo Fei Ai Za Zhi. 2012 Jun;15(6):332-9. doi: 10.3779/j.issn.1009-3419.2012.06.03. Chinese. PMID 22681919